CLINICAL TRIAL: NCT05391698
Title: Determinants of Treatment Response to State-of-the-art Interventions for Attention Deficits: Child Temperament, Cognitive Profiles and Family Dynamics
Brief Title: A Multimodal Intervention Program for Children With Attention Deficits (Child ViReal Support Program)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Crete (Other)
Responsible Party: Principal Investigator, Panagiota Dimitropoulou, Assistant Professor in Educational Psychology, University of Crete
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Neo-PRISM-C ESR-12; H2020-MSCA-ITN-2018 813546 (Other Grant/Funding Number: MARIE SKŁODOWSKA-CURIE INNOVATIVE TRAINING NETWORK (ITN))
Record Dates: First submitted 2022-05-21; First posted 2022-05-26 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Attention Deficit; Attention Deficit Disorder With Hyperactivity
Keywords: immersive virtual reality (iVR); multimodal intervention; behavioral parent training; cognitive-behavioral treatment; neurodevelopmental dysfunctions; cognitive training
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parent Training - Child Training (Group PC) (Experimental): Parents of families who will be randomized in Group PC will first take part in behavioral parent training. After the completion of the parent training program and the assessment (Time 2 assessment), their children will take part in the individualized child training program.
  Interventions: Behavioral: Behavioral Parent Training (BPT); Combination Product: Child Training (iVR + CBT)
- Child Training - Parent Training (Group CP) (Experimental): Children of families who will be randomized in Group CP will first take part in the individualized child training program. After the completion of the child training program and the assessment (Time 2 assessment), parents will take part in the behavioral parent training program.
  Interventions: Behavioral: Behavioral Parent Training (BPT); Combination Product: Child Training (iVR + CBT)

INTERVENTIONS:
Behavioral: Behavioral Parent Training (BPT) — The parent training consists of 8 weekly group sessions where parents are trained on behavior modification techniques, optimal parental practices as well as techniques for the enhancement of their children's cognitive deficits.
Combination Product: Child Training (iVR + CBT) — The child training program is comprised of 16 individualized weekly sessions. It utilizes the potentials of immersive virtual reality (iVR) technology for the training of focused and sustained attention and combines practices based on cognitive-behavioral approach for children's training on behavioral and emotional self-regulation skills.

SUMMARY:
The main aim of this study is the development and implementation of a multimodal intervention program consisting of parent training and child training which utilizes the potentials of immersive virtual reality technology (iVR) in order to test its effectiveness for children with attention deficits.

DETAILED DESCRIPTION:
Attention deficits are commonly observed in children and attention deficit hyperactivity disorder (ADHD) is one of the most commonly diagnosed childhood neurodevelopmental disorders. It is evidently known that attention deficits affect children's school, social and family life making it essential for them and their parents to receive specialized supportive services. Behavioral parent training (BPT) and cognitive-behavioral treatment (CBT) are considered evidence-based interventions for children with ADHD. In fact, they have positive effects on the management of children's behaviors, organization, reduction of parental stress and enhancement of parental self-efficacy. In addition to these traditional evidence-based interventions, immersive virtual reality (iVR) technology has been applied lately as part of intervention programs for children with attention deficits / ADHD diagnosis specifically for cognitive training.

In line with the above, investigators have designed and developed a multimodal intervention program named Child ViReal Support program. This program is comprised of parent training and child training and utilizes the potentials of iVR technology. In order to assess the efficacy of Child ViReal Support program, the investigators will conduct a randomized controlled trial, which consists of a pre-training phase, a training phase, a post-training phase and a follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Participants 9-12 years old and their parents
* ADHD diagnosis (by the approved body of Ministry of Health)
* Greek speaking participants (child and parents)
* Full Scale IQ > 80 (WISC-V) for child
* Naïve drug treatment for ADHD
* Participants able to comply with all testing and study requirements

Exclusion Criteria:

* Treatment with psychostimulants or other psychotropic drugs
* Children who received intervention based on CBT or parents who attended other behavior parent training programs
* History of comorbid neurological disorders, seizure disorder, autism spectrum disorders, psychosis, or severe dysregulation disorders that may interfere with study participation or use of virtual reality equipment
* Participants presenting a hearing or vision impairment that does not allow the tasks to be performed with the use virtual reality equipment
* Intellectual disability or WISC-V full scale IQ < 78 (1.5 standard deviations (SD) below mean)
* Non-Greek speaking child or parent
* Parents or children who refuse to give written consent for their participation in the study

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
ADHD Rating Scale-IV (ADHD-RS-IV) - Greek | 8-16 weeks
  ADHD Rating Scale-IV (Greek version, parent report) is a clinician-administered questionnaire completed by the child's parents. The scale consists of 18 questions that assess inattention (9 items) and hyperactivity/impulsivity (9 items). The total score is obtained by adding the raw scores of Inattention subscale and Hyperactivity/impulsivity subscale. Each item is rated on a 4-point Likert scale (0=Never or Rarely, 1=Sometimes, 2=Often, 3=Very Often) with total scores ranging from 0-54, while inattention subscale score and hyperactivity/impulsivity subscale score range from 0-27 each. A higher score indicates more severe ADHD symptoms.
  Changes in scores of Inattention subscale, Hyperactivity/Impulsivity subscale and Total Score will be evaluated before, during and after the intervention as well as at a follow-up assessment (3-4 months after the end of the intervention program).
Attention Network Task | 8-16 weeks
  Attention Network Task (ANT child version) is a computerized task that was developed to measure the three networks of attention in children as described by Posner and colleagues, namely the alerting network, the orienting network and the executive control network.
  The scores for each network are obtained by reaction time subtractions of different stimulus combinations (cues, congruent conditions, incongruent conditions).
  Changes in scores of alerting network, orienting network and executive control network will be evaluated before, during and after the intervention as well as at a follow-up assessment (3-4 months after the end of the intervention program).
Go/ No-Go Task | 8-16 weeks
  Go/No-Go task is a computerized task that was developed to measure attention and response inhibition. The task was developed by the research team in accordance with Conner's CPT-III task and the participant responds to certain stimuli (Go-trials) and withhold response to other stimuli (No-Go trials). There are 6 blocks of 60 trials (80% go-trials, 20% no-go trials) and there are four scores obtained from participants' responses: 1) Correct hits rate, 2) Omission error rate (do not respond in a target, inattention), 3) Commission error rate (response on a no-go trial, impulsivity) and 4) Reaction time of response on a go-trial (slower RT shows inattention).
  Changes in: 1) average correct hits rate, 2) average number of omission errors, 3) average number of commission errors and 4) reaction time variability will be evaluated before, during and after the intervention as well as at a follow-up assessment (3-4 months after the end of the intervention program).
Psychosocial Adjustment Test (Child report) | 8-16 weeks
  Psychosocial Adjustment Test is an assessment tool for the timely detection of children's skills or deficiencies in the social and emotional areas of their lives, in school adaptation as well as for the detection of difficulties in intrapersonal or interpersonal adaptation. It consists of 115 questions in a 5-point Likert scale (1=Not at all, 2=A little, 3=Moderate, 4=Very, 5=Too much) that yield five different factors: 1) Social adequacy, 2) School adequacy, 3) Emotional adequacy, 4) Self-perception and 5) Behavioral problems.
  Changes in 1) Social adequacy, 2) Emotional adequacy and 3) Behavioral problems will be evaluated before, during and after the intervention as well as at a follow-up assessment (3-4 months after the end of the intervention program).

SECONDARY OUTCOMES:
Working memory (WISC-V) | 8-16 weeks
  Working Memory Index (WISC-V) measures a child's ability to register, maintain and manipulate visual and auditory information in mind. Working Memory Index from WISC-V consists of two subscales: Digit Span and Picture Span.
  Changes in Working Memory Index results will be evaluated before, during and after the intervention as well as at a follow-up assessment (3-4 months after the end of the intervention program).
Tower of Rethymnon (similar to Tower of Hanoi or Tower of London) | 8-16 weeks
  Tower of Rethymnon is a subtest included in the Detection and Evaluation Tool for Executive Functions and it is an adaptation of the Tower of London. This test evaluates the ability to plan, to use cognitive control and to solve problems in non-verbal contexts.
  Changes in Tower of Rethymnon results will be evaluated before, during and after the intervention as well as at a follow-up assessment (3-4 months after the end of the intervention program).
Parenting Stress Index-Short Form (PSI-SF) | 8-16 weeks
  Parenting Stress Index-Short Form (PSI-SF) is a parent-report questionnaire that evaluates parenting stress, which is a variable affected by child's characteristics, parent's characteristics and by the situations surrounding their relationship. It consists of 36 items and results in five subcategories of parenting stress: 1) Parental Distress Score, 2) Parent-Child Dysfunctional Interaction Score, 3) Difficult Child Score, 4) Total Stress Score and 4) Defensive Responding Score.
  Changes in the above five scores will be evaluated before, during and after the intervention as well as at a follow-up assessment (3-4 months after the end of the intervention program).
Parenting Sense of Competence Scale (PSOC) | 8-16 weeks
  Parenting Sense of Competence Scale (PSOC) is a parent-report questionnaire that evaluates the parents' sense and perception regarding their parental ability and adequacy. It consists of 17 items and results in a Total PSOC Score. Higher score indicates greater sense of parental adequacy.
  Changes in Total PSOC Score will be evaluated before, during and after the intervention as well as at a follow-up assessment (3-4 months after the end of the intervention program).

CONTACTS AND LOCATIONS:
Overall Officials: Panagiota Dimitropoulou, PhD, Principal Investigator — University of Crete
Locations (1):
- University of Crete, Department of Psychology, Rethymno, Greece

IPD SHARING:
Plan to Share IPD: Undecided